CLINICAL TRIAL: NCT02750111
Title: Continuous Glucose Monitoring During Intecorse in Young Adults With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Orit Hamiel (Other Government)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Orit Hamiel, Head department of Pediatric Endocrinology, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Other Study IDs: 2942.1
Record Dates: First submitted 2016-04-18; First posted 2016-04-25 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Determine the incidence of hypoglycemia during / after sexual intercourse among young adults with type 1 diabetes using continuous -type sugar meter IPRO for a week.

DETAILED DESCRIPTION:
Determine the incidence of hypoglycemia during / after sexual intercourse among young adults with type 1 diabetes using continuous -type sugar meter IPRO for a week.

ELIGIBILITY:
Inclusion Criteria:

type 1 diabetes

Exclusion Criteria:

type 2 diabetes other concomitant disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05-08 (Estimated); Study Completion 2018-05-08 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | week
  Continuous glucose monitor for a week

CONTACTS AND LOCATIONS:
Overall Officials: Orit Hamiel, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes